CLINICAL TRIAL: NCT01035502
Title: A Phase II Study of Elacytarabine (CP-4055) Plus Idarubicin as Second Course Remission-Induction Therapy in Patients With Acute Myeloid Leukaemia
Brief Title: A Study of Elacytarabine (CP-4055) Plus Idarubicin as Second Course Remission-Induction Therapy in Patients With Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Collaborators: Theradex (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-205
Record Dates: First submitted 2009-12-15; First posted 2009-12-18 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Cancer; CP-4055; elacytarabine; combination; idarubicin; Acute myeloid leukaemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — 5'-oleoyl cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elacytarabine plus idarubicin (Experimental)
  Interventions: Drug: Elacytarabine plus idarubicin

INTERVENTIONS:
Drug: Elacytarabine plus idarubicin — Elacytarabine 1000 mg/m2/d will be administered as a continuous intravenous infusion (CIV) in a d 1-5 q3w cycle.
  Idarubicin will be administered IV at a fixed dose of 12 mg/ m2/d IV on d 1-3 q3w.
  It is intended that patients receive remission-induction treatment either as two combination courses, elacytarabine 1000 mg/m2/d + idarubicin 12 mg/m2/d or one combination course, elacytarabine 1000 mg/m2/d + idarubicin 12 mg/m2/d followed by one course elacytarabine 2000 mg/m2/d single therapy.

SUMMARY:
The main objective of this study is to assess the biological activity of elacytarabine in combination with idarubicin in patients with acute myeloid leukaemia who has failed the first course of a remission-induction treatment with cytarabine (ara-C). In addition, the correlation between hENT1 (human equilibrative nucleoside transporter 1) and overall survival will be studied.

DETAILED DESCRIPTION:
Elacytarabine (CP-4055) is a pro-drug of ara-C currently used in the treatment of patients with acute myeloid leukaemia. Patients with nucleoside transporter deficiency (hENT1) seem to have less benefit from cytarabine compared to those with a high expression of the transporter. Preclinical studies indicate that elacytarabine is independent of this transporter. Therefore, patients with low expression of hENT1 and treated with elacytarabine are anticipated to have a better outcome compared to patients treated with ara-C. The main objective of this study is to assess the biological activity of elacytarabine in combination with idarubicin in patients with acute myeloid leukaemia. In addition, the correlation between hENT1 (human equilibrative nucleoside transporter 1) and overall survival will be studied. Patients will be treated with elacytarabine plus idarubicin independent of their hENT1 status. Determination of the patients' hENT1 expression level will be done retrospectively. This study will also explore the safety profile of elacytarabine in combination with idarubicin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of AML according to WHO classification (excluding acute promyelocytic leukaemia)
2. Patients who have received one previous standard dose ara-C-containing regimen aiming at induction of complete remission (CR) and who have more than 5 % remaining blast cells in bone marrow following the first course of remission-induction or by other means documented residual disease (i.e. circulating blasts, persistent chloromas, other evident disease from day 12 on).
3. Patients from whom samples for determination of hENT1 status on leukemic blast cells can be taken and prepared at diagnosis and/or at baseline
4. Patients must be 18 years of age or older
5. Patients must have ECOG performance status (PS) of 0 - 2
6. Left ventricular ejection fraction (LVEF) must be >= 45 % as measured by MUGA scan or 2D ECHO within 14 days prior to start of therapy.
7. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study
8. Male and female patients must use acceptable contraceptive methods for the duration of time on study, and males also for 3 months after the last elacytarabine dose
9. Patients must be capable of understanding and complying with parameters as outlined in the protocol, and able and willing to sign a written informed consent form
10. Patients must have the following clinical laboratory values:

    * Serum creatinine <= 1.5 x the institutional upper limit of normal (ULN)
    * Total bilirubin <= 1.5 x the ULN according to national prescribing information unless considered due to Gilbert's syndrome
    * Alanine aminotransferase (ALT) (SGPT), or aspartate aminotransferase (AST) (SGOT) <= 2.5 x the ULN unless considered due to organ leukemic involvement
11. Patients must be eligible for administration of idarubicin according to current national prescribing information for idarubicin

Exclusion Criteria:

1. A history of allergic reactions to egg, idarubicin and/or other anthracyclines or other components of the products. A history of allergic reactions to ara-C of CTCAE grade 3 or 4
2. Persistent clinically significant and relevant toxicities from the previous course of chemotherapy
3. A cancer history, that according to the investigator might confound the assessment of the study endpoints
4. Patients with prior treatment with a cumulative dose of doxorubicin or equivalent exceeding 300 mg/m2 according to the following calculation index: X/300 + Y/160 < 1 where X is the doxorubicin or equivalent dose in mg/m2 and Y is the mitoxantrone dose in mg/m2. These calculations are to be used as guidance as there is no maximum cumulative dose defined in the summary of product characteristics (SPC) for idarubicin. The patient should tolerate minimum one course of combination therapy
5. Active heart disease including myocardial infarction within the previous 3 months, symptomatic coronary disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure. Any NYHA grade 3 or 4
6. Known positive status for human immunodeficiency virus (HIV)
7. Pregnant and nursing patients are excluded because the effects of elacytarabine on a fetus or a nursing child are unknown
8. Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, or psychiatric illness/social situations that may reduce compliance with study requirements
9. Patients receiving hydroxyurea within the last 12 hours prior to treatment on this protocol or any other investigational or standard cytotoxic treatment within the last 14 days, except the first remission-induction course
10. Any medical condition, which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine the rate of complete remission (CR), including complete remission with incomplete blood count recovery (CRi) in patients with AML who have not attained blast clearance after the first course of a ara-C based remission-induction therapy. | Day 21 in each course

SECONDARY OUTCOMES:
Obtain indication on the independence between hENT1 expression level and CR or CRi. Obtain guidance on disease free survival (DFS). Obtain guidance on event free survival (EFS). Characterize the safety profile of elacytarabine plus idarubicin. | Day 21 in each course
Duration of disease free survival (DFS), defined as time from CR + CRi to relapse | Study end
Duration of event free survival (EFS), defined as time from day one of therapy until relapse or death from any cause | Study end
Characterize the safety profile of elacytarabine plus idarubicin in this patient population | Study end

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University Medical Center, Durham, NC, USA
Locations (8):
- Duke University Medical Center, Durham, North Carolina, United States
- France (3):
  - CHU Lyon, Hospital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Toulouse, Hospital Purpan, Toulouse
- Germany (3):
  - Charite University Hospital Benjamin Franklin, Berlin
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Haukeland University Hospital, Bergen, Norway